CLINICAL TRIAL: NCT07235189
Title: A Randomized, Single-Center, Open-Label, Single-Dose, 4-Period, 2-Sequence, Fully Replicate Crossover Study To Assess The Bioequivalence Of A Test Fixed Dose Combination Product Versus The Co-Administered Individual Reference Products Containing Bempedoic Acid 180 MG, Ezetimibe 10 mg And Atorvastatin 40 mg In Healthy Participants
Brief Title: A Study Evaluating Bioequivalence of a Fixed Dose Combination Versus Individual Tablets of Bempedoic Acid, Ezetimibe, and Atorvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DSE-BMP-0001-CIS-MA; 2024-519849-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects
Keywords: Healthy Subjects; Bioequivalence
MeSH Terms: interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Formulation (Experimental): Healthy participants who are randomized to receive the fixed dose triplet combination with bempedoic acid 180 mg/ezetimibe 10 mg/atorvastatin 40 mg (test formulation).
  Interventions: Drug: Bempedoic acid; Drug: Ezetimibe; Drug: Atorvastatin
- Reference Formulation (Active Comparator): Healthy participants who are randomized to receive co-administration of bempedoic acid 180 mg + ezetimibe 10 mg + atorvastatin 40 mg (reference formulation).
  Interventions: Drug: Bempedoic acid; Drug: Ezetimibe; Drug: Atorvastatin

INTERVENTIONS:
Drug: Bempedoic acid — 180 mg film coated tablet administered individually or as FDC
  (Component of FDC)
  Other Names: Nilemdo®
Drug: Ezetimibe — 10 mg tablet administered individually or as FDC
  (Component of FDC)
  Other Names: Ezetrol®
Drug: Atorvastatin — 40 mg tablet administered individually or as FDC
  (Component of FDC)
  Other Names: Sortis®

SUMMARY:
Monotherapies for lowering LDL-C often do not achieve target lipid levels because they act on a single pathway, which may be insufficient in patients with high cardiovascular risk or complex lipid profiles. Triple combination therapies, targeting multiple mechanisms of cholesterol metabolism simultaneously, have demonstrated superior LDL-C reduction and better achievement of guideline recommended LDL-C goals. Additionally, combining treatments into a single regimen can improve patient adherence and compliance, further enhancing clinical outcomes. This study will test the bioequivalence of a test fixed dose combination (FDC) vs the coadministration of individual tablets.

ELIGIBILITY:
A participant is eligible for the study if he/she fulfills all of the following inclusion criteria:

1. Healthy male and female participants ≥18 and ≤60 years, at the time of signing the informed consent.
2. Body mass index (BMI) ≥18.5 and ≤30.0 kg/m^2.
3. Female participants of childbearing potential agree to undergo pregnancy tests, and if with a non-vasectomized nor infertile male partner, agree to use an appropriate method of contraception (i.e., abstinence, hormonal, intrauterine device, bilateral tubal occlusion).
4. No clinically relevant diseases captured in medical history.
5. No clinically relevant abnormalities on physical examination.
6. No clinically relevant abnormalities on vital signs.
7. No clinically relevant abnormalities on 12-lead electrocardiogram (ECG).
8. No clinically relevant abnormalities on clinical laboratory tests.
9. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) above the upper limit of normal range (ULN).
10. Estimated renal creatinine clearance (CrCl) above the lower limit of normal range, based on creatinine clearance calculation by the Cockcroft-Gault formula and normalized to an average body surface area of 1.73 m^2.
11. Willingness to accept and comply with all study procedures and restrictions.
12. Non-smoker or ex-smoker (i.e., someone who abstained from using tobacco- or nicotine-containing products for at least 3 months prior to Screening).
13. Ability to comprehend and willingness to freely sign the informed consent.

A participant is not eligible for the study at Screening if he/she fulfills any of the exclusion criteria as specified in the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameter Area Under the Curve (AUC) | Pre-dose (t=0h), and at 0.17 hours (10 minutes), 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours (Day 2), 48 hours (Day 3), and 72 hours (Day 4) postdose
  Area under the curve (AUC) from time of dosing (t=0h) to time 72 hours (AUC72h) or AUC from time of dosing (t=0h) to the time of last measurable (non-zero) concentration (AUClast) will be assessed using noncompartmental methods.
Maximum Observed Concentration (Cmax) | Pre-dose (t=0h), and at 0.17 hours (10 minutes), 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours (Day 2), 48 hours (Day 3), and 72 hours (Day 4) postdose
  Maximum observed concentration will be assessed.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters (AUCinf) | Pre-dose (t=0h), and at 0.17 hours (10 minutes), 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours (Day 2), 48 hours (Day 3), and 72 hours (Day 4) postdose
  AUC from time of dosing (t=0h) extrapolated to infinity (AUCinf) will be assessed using noncompartmental methods.
Pharmacokinetic Parameters (AUClast/AUCinf) | Pre-dose (t=0h), and at 0.17 hours (10 minutes), 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours (Day 2), 48 hours (Day 3), and 72 hours (Day 4) postdose
  AUClast/AUCinf will be assessed using noncompartmental methods.
Pharmacokinetic Parameter Time to Reach Maximum Observed Concentration (Tmax) | Pre-dose (t=0h), and at 0.17 hours (10 minutes), 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours (Day 2), 48 hours (Day 3), and 72 hours (Day 4) postdose
  Time to reach maximum observed concentration (Tmax) will be assessed.
Pharmacokinetic Parameter Terminal Half-life (t1/2) | Pre-dose (t=0h), and at 0.17 hours (10 minutes), 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours (Day 2), 48 hours (Day 3), and 72 hours (Day 4) postdose
  Terminal half-life (t1/2) will be assessed using noncompartmental methods.
Pharmacokinetic Parameter First Order Rate Constant Associated With The Terminal Portion of the Concentration-Time Curve (Kel) | Pre-dose (t=0h), and at 0.17 hours (10 minutes), 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours (Day 2), 48 hours (Day 3), and 72 hours (Day 4) postdose
  First order rate constant associated with the terminal portion of the concentration-time curve (Kel) was assessed using noncompartmental methods.
Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs) | Baseline to end of study, approximately 82 days
  AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No